CLINICAL TRIAL: NCT01276912
Title: A Multicenter, Randomized, Controlled Trial to Prevent Diabetes With Short-term Insulin Glargine Treatment or Lifestyle Intervention
Brief Title: Study TO Prevent Diabetes With Short-term Insulin Glargine Only
Acronym: STOP-GO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Jin-Kui Yang/Professor, Department of Endocrinology, Beijing Tongren Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STOP-GO-2010
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Insulin glargine — Insulin glargine therapy with a dosage adjusted to get FBG ≤ 5.3mmol / L as the goal, accompanied with a lifestyle counseling.
Behavioral: Lifestyle counseling — To give lifestyle guidance, specifically including low fat, low saturated fatty acids, rich in dietary fiber, salt restriction, limit alcohol diet plan to reduce the 5% to 10% of body weight, and to ensure a regular moderate physical activity at least 150 minutes per week.

SUMMARY:
* Pre-diabetes is a significant risk factor for the development of type 2 diabetes, as well as macrovascular and microvascular complication.
* Previous studies show that 50% or more loss in islet B-cell function even in Pre-diabetes phase. The early insulin therapy in pre-diabetes may be a strategy in preventing metabolic disorders and cardiovascular disease.
* The objective of this study is to find if an initial insulin glargine intervention in pre-diabetes (IGT and /or IFG) could be a strategy in preventing type 2 Diabetes.
* Pre-diabetes subjects will receive a insulin glargine therapy with a dosage adjusted to get FBG ≤ 5.3mmol / L as the goal. Insulin glargine treatment will be maintained for three months thereafter to find if it can prevent diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. All participants are voluntary and write informed consent 2 weeks before enrollment.
2. Fasting Blood Glucose between >= 5.6mmol/L and <7.0mmol/L, and HbA1c between >= 5.7% and <6.5%.
3. Both male and female aged between >= 25 and ≤ 65 years.
4. Participants have the ability to use self-monitoring devices to measure their blood glucose level and practice self-insulin injection.
5. Have the ability and willingness to complete the study logs and questionnaires.
6. Pregnancy test of all child-bearing age women should be negative, and they agree to adopt contraceptive measures in the study process.

Exclusion Criteria:

1. With previous diagnosis of diabetes or application of hypoglycemic drugs.
2. Preliminary screen for fasting plasma glucose lever ≥7.0mmol/L or <5.6mmol/L.
3. Preliminary screen for HbA1c result HbA1c<5.7% or ≥ 6.5%.
4. Receiving cancer treatment in the past 5 years.
5. Preliminary diagnostic anti-HIV test result positive, with no serological testing.
6. People with active tuberculosis.
7. Persons hospitalized for heart disease and received the treatment measures (such as coronary artery bypass graft CABG, percutaneous transluminal coronary angioplasty PTCA), while not include diagnostic measures (such as percutaneous coronary angiography) in the past 6 months.
8. Cardiac function evaluated by New York Heart Association criteria (NYHA) ≥ 3 cardiac function level
9. Uncontrolled high blood pressure - systolic blood pressure > 180mmHg or diastolic blood pressure > 105mmHg after treatment.
10. Stroke or transient ischemic attack episode in the past 6 months.
11. With chronic hepatitis or active liver disease, or serum AST or ALT 2.5 times the upper limit of normal.
12. Male serum creatinine ≥ 124μmol/L (1.4mg/dL); Female serum creatinine ≥ 115μmol/L (1.3mg/dL).
13. Systemic glucocorticoids applications, but other than local, eye, and inhalation applications.
14. Anemia: male hematocrit <36.0%; female <33.0%.
15. Other chronic diseases which may lead to the expected life less than 6 years or conditions that may affect life expectancy.
16. Mental disorder history.
17. Alcohol consumption (average 50g or more high spirits drink or 100g or more low spirits drink) or drug abuse.
18. Unable or unwilling to sign informed consent.
19. Cannot communicate or contact with the clinical staff.
20. Unwilling to receive insulin injection therapy or conduct self-monitoring of blood glucose.
21. Unsatisfied control of thyroid disease - subjects who are suffering thyroid disease or receiving anti-thyroid drugs or thyroid hormone treatment, show the sensitive TSH abnormalities (except for patients with low TSH who have the history of thyroid tumor or thyroid cancer receiving the inhibitor treatment).
22. Any other factors that may affect compliance or adverse events reported during the research program.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2420 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c >= 6.5% | Two years

SECONDARY OUTCOMES:
FPG >= 7.0 for two times in a month. | Two years
HbA1c >= 7.0% | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, China